CLINICAL TRIAL: NCT00530036
Title: Burden of Urinary Incontinence in Home Care Patients in the State of Geneva
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Other Study IDs: CER 06-298
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-08

CONDITIONS: Urinary Incontinence
Keywords: Mortality; Patient readmission; Institutionalization
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Continent: 54% of 699 patients followed as outpatient by the "Fondation des Services d'Aide et de Soins à Domicile" in Geneva without urinary incontinence
- Incontinent: 46% of 699 patients followed by the "Fondation des Services d'Aide et de Soins à Domicile" in Geneva and with an urinary incontinence

SUMMARY:
Urinary incontinence (UI) is a frequent problem in community-dwelling older adults and has a huge burden on health complications and healthcare costs. Although effective treatments exist, UI is frequently neglected resulting in unmet needs for continence treatment and potential negative health outcomes. The impact of UI in older patients receiving home care services has not been extensively explored. In a recent study we observed that UI was identified in 46% of 699 patients followed by the "Fondation des Services d'Aide et de Soins à Domicile" in Geneva but the impact of UI on outcome such as institutionalization, hospitalization or death is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Between July 2004 and December 2004
* 699 adults patients followed by the "Fondation des Services d'Aide et de Soins à Domicile" in Geneva (two region in the state of Geneva: Meyrin and St-Jean)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2004-01; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Jung, MD, Principal Investigator — University Hospital of Geneva (HUG)

REFERENCES:
- [Background] Jung M, Faltin DL, Rutschmann O. [Impact of urinary incontinence in community-dwelling women]. Rev Med Suisse. 2006 Oct 18;2(83):2332-5. French. PMID 17112083